CLINICAL TRIAL: NCT01128218
Title: A Phase 1 and 2 Study of 5-aminolevulinic Acid (5-ALA) to Enhance Visualisation and Resection of Malignant Glial Tumors of the Brain
Brief Title: A Study of the Specificity and Sensitivity of 5- Aminolevulinic Acid (ALA) Fluorescence in Malignant Brain Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Southern Illinois University (Other)
Collaborators: DUSA Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: COZ-SIU 10-002-1
Record Dates: First submitted 2010-05-13; First posted 2010-05-21 (Estimated); Results first posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Brain Neoplasms
Keywords: Brain Neoplasms; 5-ALA; Aminolevulinic acid; Fluorescence; Gliomas; Glioblastoma; Surgery
MeSH Terms: conditions — Brain Neoplasms; Glioma; Glioblastoma | interventions — Aminolevulinic Acid

STUDY DESIGN:
Intervention Model Description: Dose escalation study
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Phase 1 Dose Level 1 (10mg/kg) (Experimental): Dose Level 1: Participants were given a one-time, single-dose administration of oral 10mg/kg Aminolevulinic Acid (5-ALA)
  Interventions: Drug: Tumor fluorescence
- Phase 1 Dose Level 2 (20mg/kg) (Experimental): Dose Level 2: Participants were given a one-time, single-dose administration of oral 20mg/kg Aminolevulinic Acid (5-ALA)
  Interventions: Drug: Tumor fluorescence
- Phase 1 Dose level 3 (30mg/kg) (Experimental): Dose Level 3: Participants were given a one-time, single-dose administration of oral 30mg/kg Aminolevulinic Acid (5-ALA)
  Interventions: Drug: Tumor fluorescence
- Phase 1 Dose level 4 (40mg/kg) (Experimental): Dose Level 4: Participants were given a one-time, single-dose administration of oral 40mg/kg Aminolevulinic Acid (5-ALA)
  Interventions: Drug: Tumor fluorescence
- Phase 1 Dose level 5 (50mg/kg) (Experimental): Dose Level 5: Participants were given a one-time, single-dose administration of 50mg/kg Aminolevulinic Acid (5-ALA)
  Interventions: Drug: Tumor fluorescence
- Phase 2 (40mg/kg) (Experimental): Phase 2: Participants were given a one-time, single-dose administration of 40mg/kg Aminolevulinic Acid (5-ALA)
  Interventions: Drug: Tumor fluorescence

INTERVENTIONS:
Drug: Tumor fluorescence — Oral doses in phase 1 study of 10mg/kg, 20 mg/kg, 30 mg/kg, 40 mg/kg and 50 mg/kg.
  Recommended oral dose of phase 1 will be used in phase 2
  Other Names: 5-ALA; 5-aminolevulinic acid

SUMMARY:
Extent of resection is a very important prognostic factor affecting survival in individuals diagnosed with a malignant glioma. However, the infiltrative nature of the malignant glioma tumor cells produces indistinct borders between normal and malignant tissues, and the lack of easily identifiable tumor margins confounds attempts at total resection. The investigators propose to identify the borders of malignant gliomas intraoperatively using oral 5-aminolevulinic Acid (5-ALA) which results in fluorescence of the malignant cells and thereby provide an opportunity for more complete tumor resection.

When exogenous 5-ALA is provided at increased concentration the tumor cells will become fluorescent under ultraviolet light. This feature identifies the tumor cells intraoperatively and facilitates complete resection.

Data collection will include measurement of dose-limiting toxicity, tumor fluorescence, and tumor density. Data analysis will evaluate toxicity, sensitivity, and specificity of 5-ALA.

Following completion of the phase 1 portion of this trial, an additional 14 subjects will be entered at the recommended phase 2 dose level in order to further define the above parameters at the recommended phase 2 dose level.

DETAILED DESCRIPTION:
Specific Aims:

This study is intended to investigate the utility, safety and efficacy of 5-aminolevulinic acid (5-ALA) induced brain tumor fluorescence during malignant brain tumor resection. Specifically this study is intended to:

Establish a safe dose for oral 5-ALA administration. Determine the sensitivity and specificity of 5-ALA mediated fluorescence for malignant glioma tissue in the brain.

Background and Significance:

There is a considerable body of literature that suggests that completeness of resection is a positive factor for longer term survival in individuals with malignant glioma. Unfortunately, it is often difficult to completely remove a malignant brain tumor because during surgery it is sometimes very difficult to distinguish tumor from normal brain. It would be very helpful if there would be some way to help the surgeon make this distinction. Malignant glioma tumor cells (more so than normal cells) contain the biosynthetic pathways to produce protoporphyrin from a naturally occurring amino acid, 5-aminolevulinic acid (5-ALA). Protoporphyrin is the immediate precursor to hemoglobin (it is hemoglobin without the iron atom) and is fluorescent under blue light. When exogenous 5-ALA is provided at increased concentration, protoporphyrin concentration in the malignant cell increases at a rate far greater than normal brain cells and renders the malignant cell fluorescent red under blue light. This feature distinguishes the tumor cells from normal cells intraoperatively and facilitates complete resection.

Recent studies in Germany have confirmed the utility of pre-operative oral 5-ALA and intraoperative brain tumor fluorescence in aiding the resection of brain tumors in individuals with malignant brain tumors. These studies have led to oral 5-ALA to be approved for this indication by the European Medicines Agency, but oral 5-ALA has not been approved for this indication by the United States FDA. This proposal is a phase 1 and phase 2 trial that will hopefully lead to FDA approval of oral 5-ALA for intra-operative visualization of malignant brain tumors.

Experimental Plan and Methods:

In the phase 1 part of this proposed study, a minimum of 3 to a maximum of 19 patients will be administered oral 5-ALA 4 hours prior to surgery in cohorts of 3 at five escalating doses of 5-ALA (10, 20, 30, 40, or 50 mg/kg).

The following data will be collected:

* Dose-limiting toxicity data; i.e., nausea, vomiting, liver function, photo-sensitivity
* Tumor fluorescence assessed by neurosurgeon
* Tumor density from biopsies obtained by the neurosurgeon in will be assessed by neuropathology (Solid tumor, Tumor mixed infiltrating normal brain, No tumor)

This trial will evaluate:

* single dose toxicity of oral 5-ALA given pre-operatively;
* sensitivity and specificity of 5-ALA - Protoporphyrin IX (Pp IX) as an intraoperative fluorescent detection agent and aid for resection of tumor tissue remaining in the walls of the resection cavity of primary and recurrent malignant brain tumors;

Following completion of the phase 1 portion of this trial, an additional 14 subjects will be entered at the recommended phase 2 dose level in order to further define the above parameters at the recommended phase 2 dose level.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have clinically documented primary brain tumor for which resection is clinically indicated.
* Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of 5-ALA in patients <18 years of age, children are excluded from this study but will be eligible for future pediatric phase 1 single-agent trials
* ECOG (Eastern Cooperative Oncology Group) performance status <2 (Karnofsky >60%)
* Normal organ and marrow function as defined below:

  * Leukocytes > 3,000/mcL (microliter)
  * Absolute neutrophil count > 1,500/mcL
  * Platelets > 100,000/mcL
  * Total bilirubin within normal institutional limits AST (aspartate aminotransferase) (SGOT)/ALT (alanine transaminase) (SGPT) < 2.5 X institutional upper limit of normal
  * Creatinine within normal institutional limits OR Creatinine clearance > 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Agreement by women of child-bearing potential and men to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients may not be receiving any other investigational agents at the time of entry into the study
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 5-ALA
* Personal or family history of porphyrias
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because 5-ALA is of unknown teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with 5-ALA, breastfeeding should be discontinued if the mother is treated with 5-ALA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2021-02 (Actual); Study Completion 2021-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey W Cozzens, MD, Principal Investigator — Southern Illinois University School of Medicine
Locations (1):
- Southern Illinois University School of Medicine, Springfield, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keles GE, Anderson B, Berger MS. The effect of extent of resection on time to tumor progression and survival in patients with glioblastoma multiforme of the cerebral hemisphere. Surg Neurol. 1999 Oct;52(4):371-9. doi: 10.1016/s0090-3019(99)00103-2. PMID 10555843
- [Background] Sanai N, Berger MS. Glioma extent of resection and its impact on patient outcome. Neurosurgery. 2008 Apr;62(4):753-64; discussion 264-6. doi: 10.1227/01.neu.0000318159.21731.cf. PMID 18496181
- [Background] Stummer W, Pichlmeier U, Meinel T, Wiestler OD, Zanella F, Reulen HJ; ALA-Glioma Study Group. Fluorescence-guided surgery with 5-aminolevulinic acid for resection of malignant glioma: a randomised controlled multicentre phase III trial. Lancet Oncol. 2006 May;7(5):392-401. doi: 10.1016/S1470-2045(06)70665-9. PMID 16648043
- [Background] Tonn JC, Stummer W. Fluorescence-guided resection of malignant gliomas using 5-aminolevulinic acid: practical use, risks, and pitfalls. Clin Neurosurg. 2008;55:20-6. No abstract available. PMID 19248665
- [Derived] Cozzens JW, Lokaitis BC, Delfino K, Hoeft A, Moore BE, Fifer AS, Amin DV, Espinosa JA, Jones BA, Acakpo-Satchivi L. A Phase 2 Sensitivity and Selectivity Study of High-Dose 5-Aminolevulinic Acid in Adult Patients Undergoing Resection of a Newly Diagnosed or Recurrent Glioblastoma. Oper Neurosurg. 2024 Nov 11;29(1):71-79. doi: 10.1227/ons.0000000000001417. PMID 39526779
- See also: Brain Cancer — http://www.nlm.nih.gov/medlineplus/braincancer.html
- See also: Cancer — http://www.nlm.nih.gov/medlineplus/cancer.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 Dose Level 1 (10mg/kg): Dose Level 1: Participants were given a one-time, single-dose administration of oral10mg/kg Aminolevulinic Acid (5-ALA)
- Phase 1 Dose Level 5 (50mg/kg): Dose Level 5: Participants were given a one-time, single-dose administration of oral 50mg/kg Aminolevulinic Acid (5-ALA)
- Phase 2 (40mg/kg): Phase 2 (40mg/kg): Participants were given a one-time, single-dose administration of oral 50mg/kg Aminolevulinic Acid (5-ALA)
Period: Overall Study
Arm/Group | Phase 1 Dose Level 1 (10mg/kg) | Phase 1 Dose Level 2 (20mg/kg) | Phase 1 Dose Level 3 (30mg/kg) | Phase 1 Dose Level 4 (40mg/kg) | Phase 1 Dose Level 5 (50mg/kg) | Phase 2 (40mg/kg)
Started | 3 | 3 | 3 | 4 | 6 | 14
Completed | 3 | 3 | 3 | 4 | 6 | 14
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 1 Dose Level 1 (10mg/kg): Phase 1 Dose Level 1: Participants were given a one-time, single-dose administration of oral 10mg/kg Aminolevulinic Acid (5-ALA)
- Phase 1 Dose Level 2 (2omg/kg): Phase 1 Dose Level 2: Participants were given a one-time, single-dose administration of oral 20mg/kg Aminolevulinic Acid (5-ALA)
- Phase 1 Dose Level 3 (30mg/kg): Phase 1 Dose Level 3: Participants were given a one-time, single-dose administration of oral 30mg/kg Aminolevulinic Acid (5-ALA)
- Phase 1 Dose Level 4 (40mg/kg): Phase 1 Dose Level 4: Participants were given a one-time, single-dose administration of oral 40mg/kg Aminolevulinic Acid (5-ALA)
- Phase 1 Dose Level 5 (50mg/kg): Phase 1 Dose Level 1: Participants were given a one-time, single-dose administration of oral 50mg/kg Aminolevulinic Acid (5-ALA)
- Phase 2 (40mg/kg): Phase 2: Participants were given a one-time, single-dose administration of oral 40mg/kg Aminolevulinic Acid (5-ALA)
- Total: Total of all reporting groups
Arm/Group | Phase 1 Dose Level 1 (10mg/kg) | Phase 1 Dose Level 2 (2omg/kg) | Phase 1 Dose Level 3 (30mg/kg) | Phase 1 Dose Level 4 (40mg/kg) | Phase 1 Dose Level 5 (50mg/kg) | Phase 2 (40mg/kg) | Total
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 6 | 14 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3 | 1 | 6 | 6 | 19
  >=65 years | 2 | 1 | 0 | 3 | 0 | 8 | 14
Age, Continuous [Mean (Full Range); unit: years] | 64 [32 to 87] | 61 [54 to 74] | 63 [62 to 67] | 71 [63 to 77] | 52.5 [44 to 62] | 56.36 [21 to 84] | 58.63 [21 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 0 | 1 | 3 | 8 | 16
  Male | 0 | 2 | 3 | 3 | 3 | 6 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 3 | 3 | 3 | 3 | 6 | 14 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 1
  White | 3 | 2 | 3 | 4 | 6 | 14 | 32
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 4 | 6 | 14 | 33

OUTCOME MEASURES:

1. Primary Outcome: Establish a Safe Dose for Oral 5-ALA Administration
Description: Dose escalation from 10mg/kg to 50mg/kg to determine optimal 5-ALA dose
Time Frame: 6 months
Population: There were no dose limiting toxicities observed at any dose level arm. Therefore, the 40mg/kg dose was arbitrarily chosen for the phase 2 portion of the study.
Measure: Number; unit: Dose Limiting Toxicity
Groups:
- Phase 1 Dose Level 2 (20mg/kg): Phase 1 Dose Level 2: Participants were given a one-time, single-dose administration of oral 20mg/kg Aminolevulinic Acid (5-ALA)
- Phase 1 Dose Level 5 (50mg/kg): Phase 1 Dose Level 5: Participants were given a one-time, single-dose administration of oral 50mg/kg Aminolevulinic Acid (5-ALA)
Arm/Group | Phase 1 Dose Level 1 (10mg/kg) | Phase 1 Dose Level 2 (20mg/kg) | Phase 1 Dose Level 3 (30mg/kg) | Phase 1 Dose Level 4 (40mg/kg) | Phase 1 Dose Level 5 (50mg/kg)
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 6
Dose Limiting Toxicity | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Determine the Sensitivity, Specificity, and Positive Predictive Value of 5-ALA Mediated Fluorescence for Malignant Glioma Tissue in the Brain.
Description: The neurosurgeon will take two small biopsies per patient from areas identified as obvious tumor and areas in the wall of the resection cavity that were judged to be normal, non-eloquent brain. A neuropathologist will review all biopsy specimens, including those taken from the solid tumor. Pathologic confirmation of tumor type will be made by the study reference neuropathologist.
  We assessed 5-ALA's resulting fluorescence for distinguishing tumor within the brain, where
  True Positive: Fluorescence showing Tumor and Biopsy result Tumor False Positive: Fluorescence showing Tumor and Biopsy result No Tumor True Negative: No Fluorescence and Biopsy result No Tumor False Negative: No Fluorescence and Biopsy result Tumor
  These values represent the characteristics of 5-ALA aka its ability to distinguish tumor from non-tumor. From these parameters we determined sensitivity, specificity and the positive and negative predictive values.
Time Frame: Baseline
Population: Assessing sensitivity, specificity, positive predictive value, and negative predictive value in Phase 2 Study Population of N=14 Patients at 40 mg/kg Dose
Measure: Number; unit: Percentage
Units Other Than Participants: Biopsies
Groups:
- Phase 2 Dose Level 1 (40mg/kg): A single arm in this open-label study where all patients are treated with the study drug - 5-aminolevulinic acid. Areas of the brain that are fluorescent and areas that are not fluorescent are evaluated for presence of tumor cells
  Tumor fluorescence: Oral Phase 2 dose: 40mg/kg.
Arm/Group | Phase 2 Dose Level 1 (40mg/kg)
Number analyzed (Participants) | 14
Number analyzed (Biopsies) | 28
Percentage
  Sensitivity | 63.64
  Specificity | 100
  Positive Predictive Value | 100
  Negative Predictive Value | 42.86

3. Other Pre Specified Outcome: Assess 5-ALA's Resulting Fluorescence for Distinguishing Tumor Within the Brain
Description: Under blue light, the neurosurgeon will take two small biopsies per patient from areas identified as obvious tumor (fluorescent) and areas in the wall of the resection cavity that were judged to be normal (but possibly edematous), non-eloquent brain (non-fluorescent). A neuropathologist will review all biopsy specimens, including those taken from the solid tumor. Pathologic confirmation of tumor type will be made by the study reference neuropathologist.
  We assessed 5-ALA's resulting fluorescence for distinguishing tumor within the brain, where
  True Positive: Fluorescence showing Tumor and Biopsy result Tumor False Positive: Fluorescence showing Tumor and Biopsy result No Tumor True Negative: No Fluorescence and Biopsy result No Tumor False Negative: No Fluorescence and Biopsy result Tumor
  These values represent the characteristics of 5-ALA aka its ability to distinguish tumor from non-tumor.
Time Frame: Baseline
Population: Phase 2 Study Population of N=14 Patients at 40 mg/kg Dose
Measure: Number; unit: Biopsies
Units Other Than Participants: Biopsies
Arm/Group | Phase 2 Dose Level 1 (40mg/kg)
Number analyzed (Participants) | 14
Number analyzed (Biopsies) | 28
Biopsies
  True Positives | 14
  True Negatives | 6
  False Positives | 0
  False Negatives | 8

ADVERSE EVENTS:
Time Frame: 6 years
Groups:
- Phase 1, Dose Level 1 (10mg/kg): Phase 1 Dose Level 1: Participants were given a one-time, single-dose administration of oral 10mg/kg Aminolevulinic Acid (5-ALA)
- Phase 1, Dose Level 2 (20mg/kg): Phase 1 Dose Level 2: Participants were given a one-time, single-dose administration of oral 20mg/kg Aminolevulinic Acid (5-ALA)
- Phase 1, Dose Level 3 (30mg/kg): Phase 1 Dose Level 3: Participants were given a one-time, single-dose administration of oral 30mg/kg Aminolevulinic Acid (5-ALA)
- Phase 1, Dose Level 4 (40mg/kg): Phase 1 Dose Level 4: Participants were given a one-time, single-dose administration of oral 40mg/kg Aminolevulinic Acid (5-ALA)
- Phase 1, Dose Level 5 (50mg/kg): Phase 1 Dose Level 5: Participants were given a one-time, single-dose administration of oral 50mg/kg Aminolevulinic Acid (5-ALA)
- Phase 2 (40mg/kg): Phase 2 Dose (40mg/kg): Participants were given a one-time, single-dose administration of oral 40mg/kg Aminolevulinic Acid (5-ALA)
Arm/Group | Phase 1, Dose Level 1 (10mg/kg) | Phase 1, Dose Level 2 (20mg/kg) | Phase 1, Dose Level 3 (30mg/kg) | Phase 1, Dose Level 4 (40mg/kg) | Phase 1, Dose Level 5 (50mg/kg) | Phase 2 (40mg/kg)
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/3 | 0/3 | 0/4 | 0/6 | 0/14
Serious Adverse Events (participants affected / at risk) | 2/3 | 0/3 | 0/3 | 0/4 | 0/6 | 2/14
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/4 | 0/6 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1, Dose Level 1 (10mg/kg) (N=3) | Phase 1, Dose Level 2 (20mg/kg) (N=3) | Phase 1, Dose Level 3 (30mg/kg) (N=3) | Phase 1, Dose Level 4 (40mg/kg) (N=4) | Phase 1, Dose Level 5 (50mg/kg) (N=6) | Phase 2 (40mg/kg) (N=14)
death (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — The patient was coded secondary to the ventricular tachycardia change to ventricular fibrillation and asystole in 20 seconds.
scalp wound abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Admitted to hospital for an infected cranial wound. Subject seen by infectious disease specialist Incision and drainage of cranial wound, removal of cranial bone flap, and revision of cranial wound done.
severe cerebral edema (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — blown pupils; intubated; increased cerebral edema; evidence of increased density in the basilar subarachnoid spaces and did not show true subarachnoid hemorrhage; culture positive for Gram Negative Rods.
partial seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — "Had a partial seizure today despite Keppra prophylaxis."

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT01128218/Prot_SAP_000.pdf